CLINICAL TRIAL: NCT04786964
Title: A Randomized, Open-Label, Phase 3 Study of Cosibelimab (CK-301) in Combination With Platinum+Pemetrexed Chemotherapy in Subjects With First-Line Metastatic Non-squamous Non-Small Cell Lung Cancer
Brief Title: Study of Pemetrexed+Platinum Chemotherapy With or Without Cosibelimab in First Line Metastatic Non-squamous NSCLC
Acronym: CONTERNO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Regional political conflict
Sponsor: Checkpoint Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CK-301-301
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Non-squamous Non Small Cell Lung Cancer
Keywords: Metastatic; non-small cell lung cancer; nonsquamous; PD-L1; PD-1; PDL1; PD1; Lung neoplasms; Cosibelimab; Non-squamous NSCLC; Carcinoma, non-small cell lung; Antineoplastic agents; CK-301; Anti-PD-L1
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; Carboplatin; Pemetrexed; Folic Acid; Vitamin B 12; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cosibelimab (Experimental): Participants receive cosibelimab 1200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by cosibelimab 1200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression.
  Interventions: Drug: Cosibelimab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Dietary Supplement: Folic acid 350-1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4mg
- Control (Active Comparator): Participants receive pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin AUC 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pemetrexed 500 mg/m^2 IV Q3W until progression.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Dietary Supplement: Folic acid 350-1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4mg

INTERVENTIONS:
Drug: Cosibelimab — IV infusion
  Arms: Cosibelimab
Drug: Cisplatin — IV infusion
Drug: Carboplatin — IV infusion
Drug: Pemetrexed — IV infusion
Dietary Supplement: Folic acid 350-1000 μg — Orally; at least 5 doses of folic acid must be taken during the 7 days preceding the first dose of pemetrexed, and folic acid dosing must continue during the full course of therapy and for 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B12 1000 μg — Intramuscular injection in the week preceding the first dose of pemetrexed and once every 3 cycles thereafter. Subsequent vitamin B12 injections may be given the same day as pemetrexed administration.
Drug: Dexamethasone 4mg — For prophylaxis; orally twice per day (or equivalent). Taken the day before, day of, and day after pemetrexed administration.

SUMMARY:
This is an efficacy and safety study of cosibelimab (CK-301) combined with pemetrexed/platinum chemotherapy versus pemetrexed/platinum chemotherapy alone in participants with advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) who have not previously received systemic therapy for advanced disease. Participants will be randomly assigned in a 2:1 ratio to receive cosibelimab combined with pemetrexed/platinum (Investigators choice of cisplatin or carboplatin), OR pemetrexed/platinum (Investigators choice of cisplatin or carboplatin).

The primary hypothesis is that cosibelimab in combination with pemetrexed/platinum chemotherapy prolongs Overall Survival (OS) compared to pemetrexed/platinum chemotherapy alone.

DETAILED DESCRIPTION:
CK-301-301 is a Phase 3, open-label, multicenter, randomized, active-controlled study of the safety and efficacy of IV administered cosibelimab 1200 mg Q3W in combination with platinum/pemetrexed chemotherapy versus chemotherapy alone in subjects with NSCLC who have not previously received systemic therapy for advanced disease and in whom epidermal growth factor receptor-directed therapy or anaplastic lymphoma kinase-directed therapy was not indicated. Subjects were randomized 2:1 to receive cosibelimab 1200 mg in combination with pemetrexed and platinum therapy, or pemetrexed and platinum therapy alone. Subjects were stratified by smoking status (never versus former/current), cisplatin vs carboplatin, and PD-L1 status (Tumor Proportion Score [TPS] < 1% vs 1-49% vs ≥ 50%) prior to randomization. Subjects with unevaluable PD-L1 status were included with the TPS < 1% group.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically-confirmed or cytologically confirmed diagnosis of stage IV non-squamous NSCLC.
* Has confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated.
* Has measurable disease.
* Has not received prior systemic treatment for their advanced/metastatic NSCLC.
* Can provide tumor tissue.
* Has a life expectancy of at least 3 months.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Has adequate organ function
* If female of childbearing potential, is willing to use adequate contraception for the course of the study through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.
* If male with a female partner(s) of child-bearing potential, must agree to use adequate contraception starting with the first dose of study medication through 180 days after the last dose of study medication and chemotherapeutic agents.

Exclusion Criteria:

* Has predominantly squamous cell histology NSCLC.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to administration of study medication.
* Before the first dose of study medication: a) Has received prior systemic cytotoxic chemotherapy for metastatic disease, b) Has received antineoplastic biological therapy (e.g., erlotinib, crizotinib, cetuximab), c) Had major surgery (<3 weeks prior to first dose).
* Received radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study medication.
* Completed palliative radiotherapy within 7 days of the first dose of study medication.
* Is expected to require any other form of antineoplastic therapy while on study.
* Received a live-virus vaccination within 30 days of planned start of study medication.
* Has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, peritoneal carcinomatosis.
* Known history of prior malignancy except if participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy, except for successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb).
* Known sensitivity to any component of cisplatin, carboplatin or pemetrexed.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Is on chronic systemic steroids.
* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Is unable or unwilling to take folic acid or vitamin B12 supplementation.
* Had prior treatment with any other anti-programmed cell death-1 (PD-1), or PD-ligand 1 (PD-L1) or PD-L2 agent or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Has an active infection requiring therapy.
* Has known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or C.
* Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* Is a known regular user of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Has symptomatic ascites or pleural effusion.
* Has active or history of interstitial lung disease or a history of (non infectious) pneumonitis that required steroids or current pneumonitis.
* Has had an allogeneic tissue/solid organ transplant.
* Any known uncontrolled or significant cardiovascular disease.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Research Site, Vitória, Brazil
- Research Site, Tbilisi, Georgia
- Research Site, Kota Bharu, Malaysia
- Research Site, Wellington, New Zealand
- Research Site, Lima, Peru
- Russia (15):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Kaliningrad
  - Research Site, Kazan'
  - Research Site, Kursk
  - Research Site, Kuzmolovskiy
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Sochi
  - Research Site, Tomsk
  - Research Site, Volgograd
- Research Site, Pretoria, South Africa
- Research Site, Chiang Mai, Thailand

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized 2:1 to receive cosibelimab 1200 mg in combination with pemetrexed and platinum therapy, or pemetrexed and platinum therapy alone. The platinum therapy, cisplatin, or carboplatin was based on Investigator's choice. Subjects were stratified by smoking status (never vs former/current), cisplatin vs carboplatin, and PD-L1 status prior to randomization. Subjects with unevaluable PD-L1 status were included with the TPS < 1% group.
Period: Overall Study
Arm/Group | Cosibelimab | Control
Started | 19 | 6
Completed | 19 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 25 patients were enrolled in the study as the study was prematurely terminated due to a regional political conflict that prevented ongoing study conduct.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cosibelimab | Control | Total
Number analyzed (Participants) | 19 | 6 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 4 | 16
  >=65 years | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 12 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 6 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 19 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Defined as the time from randomization to death due to any cause.
Time Frame: Approximately 3 years.
Population: Due to the Russia/Ukraine conflict initiating during the study start up, the study was put on hold, and then the study terminated prior to efficacy analysis. This study will not be used to support marketing application approval.
Arm/Group | Cosibelimab | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Defined as the time from randomization until disease progression by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Time Frame: Approximately 3 years.
Population: as for outcome 1
Arm/Group | Cosibelimab | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Defined as the proportion of participants who have a confirmed complete response or partial response per RECIST v1.1
Time Frame: Approximately 3 years.
Population: as for outcome 1
Arm/Group | Cosibelimab | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from the earliest date of documented response until earliest date of disease progression (per RECIST v1.1) or death from any cause, whichever comes first.
Time Frame: Approximately 3 years.
Population: as for outcome 1
Arm/Group | Cosibelimab | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a study participant administered study drug and which does not necessarily have to have a causal relationship with this study drug.
Time Frame: Approximately 2 years.
Population: Adverse event monitoring was performed throughout the study; after the end of treatment, subjects were followed for a minimum of 30 days for AE monitoring through the end of the study, which was up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Cosibelimab | Control
Number analyzed (Participants) | 19 | 6
Participants | 14 | 6

ADVERSE EVENTS:
Time Frame: Adverse event monitoring was performed throughout the study; after the end of treatment, subjects were followed for a minimum of 30 days for AE monitoring and up to 90 days for SAEs and irAEs through study completion, up to 24 months. Note the study was prematurely terminated due to the geopolitical conflict in the region.
Arm/Group | Cosibelimab | Control
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/6
Other Adverse Events (participants affected / at risk) | 14/19 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cosibelimab (N=19) | Control (N=6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cosibelimab (N=19) | Control (N=6)
Asthenia (General disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 8 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 3
Decreased appetite (Gastrointestinal disorders) | 3 | 1
Other abnormal labs (Investigations) | 7 | 4
Hypothyroidism (Endocrine disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Immune-mediated thyroiditis (Endocrine disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Non-cardiac chest pain (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Type I hypersensitivity (Immune system disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Prostate calcifications (Reproductive system and breast disorders) | 0 | 1
Edema (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotonia (Musculoskeletal and connective tissue disorders) | 0 | 1
Vascular leukoencephalopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor owns and publishes clinical trial results. The PI cannot publish results unless and until requested in writing by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04786964/Prot_SAP_001.pdf